CLINICAL TRIAL: NCT06139068
Title: The Effect of Narrative Group Counseling on Psychological Resilience in Nursing Students
Brief Title: Narrative Group Counseling and Psychological Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023-208536434
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Psychological Resilience
Keywords: Psychological Resilience; Narrative Therapy; Nursing Students; Psychiatric nursing

STUDY DESIGN:
Intervention Model Description: The research was used parallel group, randomized, controlled experimental design.
Who Masked: Participant, Outcomes Assessor
Masking Description: An intervention was applied to both groups and blinding of the participants was ensured. It is planned to analyze the data by a statistician independent of the research. In the study, blinding was not possible since it was the researcher who implemented the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Narrative group counseling consists of 8 sessions and will be applied to the intervention group by the researcher.
  Interventions: Other: Narrative Group Counseling
- Control (Active Comparator): For the control group, 4 sessions stress coping interviews will be held after the information meeting, apart from the students' routine practices.
  Interventions: Other: stress coping interviews

INTERVENTIONS:
Other: Narrative Group Counseling — Two of the principles that explain how narrative therapy works are: to always maintain a stance of curiosity on the part of the practitioner and to ask questions to which the practitioner does not actually know the answers and to which the answer is known to the participants. To guide therapeutic conversations that include these questions, Michael White and David Epston have designed a series of conversation maps in the application of narrative therapy. Taking these maps into consideration, the sessions were planned with the guidance of relevant literature and structured with expert opinions. Group counseling was applied to the intervention group once a week in 8 sessions. The intervention was completed face to face, in a calm, quiet and bright environment, with a round seating plan. One session lasted 90 minutes. Each session was completed in two parts with a 10-minute break.
  Arms: intervention
Other: stress coping interviews — In addition to the students' routine practices, four sessions of stress coping interviews will be held for the control group, with an interval of two weeks, after the information meeting.
  Arms: Control

SUMMARY:
This study aims to examine the effect of narrative group counseling applied to nursing students studying at a public university on psychological resilience. The research was used parallel group, randomized, controlled experimental design. According to the power analysis results, the sample size was determined to be at least 54 people. Due to possible losses, 25% more people were included in the study and 68 students who met the inclusion criteria were assigned to the intervention (n = 34) and control group (n = 34). In the study, the assignment of students to the intervention and control groups were made by stratified randomization(gender,class). Due to the fact that nursing department courses continued all day on weekdays, limited transportation and winter conditions, students from the intervention group (n = 7) and the control group (n = 5) did not want to continue the sessions. The implementation of the research was completed with a total of 56 students, with n=27 in the intervention group and n=29 in the control group. Personal information forms and Adult Resilience Scale were used to obtain research data. The data collection process was carried out in four stages: pre-test, post-test, 3-month follow-up test and 6-month follow-up test.

DETAILED DESCRIPTION:
The intervention group received eight sessions of narrative group counseling. The control group also received four session of stress management training.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being 18 years of age or older

Exclusion Criteria:

* Having a neurological or psychiatric diagnosis based on self-report
* Having attended another similar program, individually or with a group.
* Having attended another similar program, individually or with a group, for at least 1 year ago.
* Being a foreign student.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Resilience Scale For Adults (RSA) | before the intervention
  Resilience Scale for Adults The Turkish validity and reliability of the scale developed by Fribourg et al. (2003) was conducted by Basım and Çetin (2011). The 33-item scale consists of six sub-dimensions: "Self-Perception", "Future Perception", "Structural Form", "Social Competence", "Family Cohesion" and "Social Resources".
Resilience Scale For Adults (RSA) | eight weeks after the start of intervention
  Resilience Scale for Adults The Turkish validity and reliability of the scale developed by Fribourg et al. (2003) was conducted by Basım and Çetin (2011). The 33-item scale consists of six sub-dimensions: "Self-Perception", "Future Perception", "Structural Form", "Social Competence", "Family Cohesion" and "Social Resources".
Resilience Scale For Adults (RSA) | three months after implementation of the intervention
  Resilience Scale for Adults The Turkish validity and reliability of the scale developed by Fribourg et al. (2003) was conducted by Basım and Çetin (2011). The 33-item scale consists of six sub-dimensions: "Self-Perception", "Future Perception", "Structural Form", "Social Competence", "Family Cohesion" and "Social Resources".
Resilience Scale For Adults (RSA) | six months after implementation of the intervention
  Resilience Scale for Adults The Turkish validity and reliability of the scale developed by Fribourg et al. (2003) was conducted by Basım and Çetin (2011). The 33-item scale consists of six sub-dimensions: "Self-Perception", "Future Perception", "Structural Form", "Social Competence", "Family Cohesion" and "Social Resources".

CONTACTS AND LOCATIONS:
Overall Officials: SULTAN AYAZ ALKAYA, Prof.Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)